CLINICAL TRIAL: NCT04585412
Title: A Randomized, Single-dose, Two-way Crossover Study to Evaluate Bioequivalence of Two Formulations of Palonosetron After Intravenous Administration of Palonosetron in Healthy Volunteers Under Fasting Conditions
Brief Title: Evaluate Bioequivalence of Palonosetron (0.25mg/5mL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: YSP-RLH3001-01
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Chemotherapy-induced Nausea and Vomiting, Prophylaxis
MeSH Terms: conditions — Vomiting | interventions — Palonosetron

STUDY DESIGN:
Intervention Model Description: An open-label, randomized, balanced, two-treatment, two-period, twosequence, single dose, two-way crossover study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palonosetron (Stothu®) (Experimental): Stothu® Solution for Injection 0.25 mg/5 mL
  Interventions: Drug: Palonosetron
- Palonosetron (Aloxi®) (Active Comparator): Aloxi® Solution for Injection 0.25 mg/5mL
  Interventions: Drug: Palonosetron

INTERVENTIONS:
Drug: Palonosetron — Pharmacokinetic study under fasting conditions
  Other Names: Stothu®

SUMMARY:
A randomized, single-dose, two-way crossover study to evaluate bioequivalence of two formulations of palonosetron after intravenous administration of palonosetron in healthy volunteers under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female subjects between 20-45 years of age (inclusive) at the screening visit.
2. Body mass index (BMI) between 18 and 27 kg/m2 (not inclusive) at the screening visit.
3. Acceptable medical history and physical examination including:

   * no particular clinically significant abnormalities in ECG results within six months prior to Period I dosing.
   * no particular clinical significance in general disease history within two months prior to Period I dosing.
4. Acceptable biochemistry determinations (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to Period I dosing, which includes AST (SGOT), ALT (SGPT), γ-GT, alkaline phosphatase, total bilirubin, albumin, glucose, BUN, uric acid, creatinine, total cholesterol and triglyceride (TG).
5. Acceptable hematology (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to Period I dosing, which includes hemoglobin, hematocrit, red blood cell count, white blood cell count with differentials and platelets.
6. Acceptable urinalysis (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to Period I dosing, which includes pH, blood, glucose, ketones, bilirubin and protein.
7. Female of childbearing potential practicing an acceptable method of birth control for the duration of the study.
8. Have signed the written informed consent to participate in the study.

Exclusion Criteria:

1. A clinically significant disorder involving the cardiovascular, respiratory, hepatic, renal, urinary tract, gastrointestinal, immunologic, hematologic, endocrine or neurologic system(s) or psychiatric disease.
2. A clinically significant illness or surgery within four weeks prior to Period I dosing.
3. History of gastrointestinal obstruction, inflammatory bowel disease, gallbladder disease, pancreas disorder over last two years or history of gastrointestinal tract surgery over last five years.
4. History of kidney disease or urination problem over last two years deemed by the investigator to be clinically significant.
5. Known or suspected history of drug abuse within lifetime.
6. History of alcohol addiction or abuse within last five years or use of more than 7 units of alcohol per week within two weeks prior to dosing. (1 unit of alcohol = 10 g of alcohol or about 350 mL of beer or about 83 mL of red wine or about 30 mL of beverage containing 40% (v/v) alcohol).
7. History of allergic response(s) to palonosetron or any other related drugs.
8. Evidence of chronic or acute infectious diseases.
9. Positive result for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), or human immunodeficiency virus (HIV).
10. Female subjects demonstrating a positive pregnancy screen prior to the study.
11. Female subjects who are currently breastfeeding.
12. Taking any drug known to induce or inhibit hepatic drug metabolism within four weeks prior to Period I dosing. Examples of inducers include: piperidines, carbamazepine, dexamethasone and rifampin. Examples of inhibitors include: cimetidine, diphenhydramine, fluvastatin, methadone and ranitidine.
13. Taking any prescription medications within four weeks or any nonprescription medications (excluding flu vaccination) within two weeks prior to Period I dosing.
14. Use of any investigational drug within four weeks prior to Period I dosing.
15. Donating more than 250 mL of blood within two months prior to Period I dosing or donating plasma (e.g. plasmapheresis) within two weeks prior to Period I dosing.
16. Any other medical reason as determined by the investigator.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2020-10-24 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | 0 (pre-dose), ≤2, 5, 15, and 30 minutes, and 1, 2, 4, 6, 12, 24, 48, 72, 96, 120, 144, and 168 hours post dose
  The two-sided 90% confidence interval for the difference of means in natural log-transformed Cmax, AUC0-t and AUC0-∞ between test and reference drug will be calculated.
Time to reach peak concentration (Tmax) | 0 (pre-dose), ≤2, 5, 15, and 30 minutes, and 1, 2, 4, 6, 12, 24, 48, 72, 96, 120, 144, and 168 hours post dose
  The two-sided 90% confidence interval for the difference of means in natural log-transformed Cmax, AUC0-t and AUC0-∞ between test and reference drug will be calculated.
Area under the concentration-time curve from time zero to time of last quantifiable concentration (AUC0-t) | 0 (pre-dose), ≤2, 5, 15, and 30 minutes, and 1, 2, 4, 6, 12, 24, 48, 72, 96, 120, 144, and 168 hours post dose
  The two-sided 90% confidence interval for the difference of means in natural log-transformed Cmax, AUC0-t and AUC0-∞ between test and reference drug will be calculated.
Area under the concentration-time curve from time zero to infinity (AUC0-∞) | 0 (pre-dose), ≤2, 5, 15, and 30 minutes, and 1, 2, 4, 6, 12, 24, 48, 72, 96, 120, 144, and 168 hours post dose
  The two-sided 90% confidence interval for the difference of means in natural log-transformed Cmax, AUC0-t and AUC0-∞ between test and reference drug will be calculated.
Elimination rate constant (入z) | 0 (pre-dose), ≤2, 5, 15, and 30 minutes, and 1, 2, 4, 6, 12, 24, 48, 72, 96, 120, 144, and 168 hours post dose
  The two-sided 90% confidence interval for the difference of means in natural log-transformed Cmax, AUC0-t and AUC0-∞ between test and reference drug will be calculated.
Terminal elimination half-life (t1/2) | 0 (pre-dose), ≤2, 5, 15, and 30 minutes, and 1, 2, 4, 6, 12, 24, 48, 72, 96, 120, 144, and 168 hours post dose
  The two-sided 90% confidence interval for the difference of means in natural log-transformed Cmax, AUC0-t and AUC0-∞ between test and reference drug will be calculated.
Ratio of AUC0-t to AUC0-∞ | 0 (pre-dose), ≤2, 5, 15, and 30 minutes, and 1, 2, 4, 6, 12, 24, 48, 72, 96, 120, 144, and 168 hours post dose
  The two-sided 90% confidence interval for the difference of means in natural log-transformed Cmax, AUC0-t and AUC0-∞ between test and reference drug will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan